CLINICAL TRIAL: NCT06809751
Title: Evaluating Efficacy and Safety of Oral Melatonin in Acute Central Serous Chorioretinopathy (CSCR): a Double-blind Randomized Clinical Trial
Brief Title: Evaluating Efficacy and Safety of Oral Melatonin in Acute Central Serous Chorioretinopathy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mohsen Pourazizi (Other)
Responsible Party: Sponsor-Investigator, Mohsen Pourazizi, Assistant Professor of Ophthalmology, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.ARI.MUI.REC.1403.234
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Central Serous Chorioretinopathy; Melatonin; Ocular Diseases; Visual Acuity; Macula Abnormality
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case group: treatment with oral melatonin (Experimental): In the case group, the patients with central serous chorioretinopathy will receive oral melatonin within one month and outcomes will be assessed after finishing the course of the treatment, and 1 and 3 months later.
  Interventions: Drug: melatonin 3mg
- Placebo group: treatment with placebo (Placebo Comparator): In the placebo group, the patients with central serous chorioretinopathy will receive the placebo substance after finishing the course of the treatment, and 1 and 3 months later.
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: melatonin 3mg — In this group, participants will be randomly assigned to take 3 mg tablets of melatonin twice a day for 1 month.
  Arms: Case group: treatment with oral melatonin
Drug: Placebo Drug — The placebo is also prepared in the form of tablets with similar packaging as melatonin by the pharmaceutical company. Participants will be randomly assigned to take placebo with the same frequency and duration as melatonin (twice a day for 1 month).
  Arms: Placebo group: treatment with placebo

SUMMARY:
The goal of this clinical trial is to learn if oral melatonin can enhance visual acuity and central macular thickness in central serous chorioretinopathy (CSCR) in adults. The main questions it aims to answer are:

1. How does melatonin affect central macula thickness in CSCR?
2. How does melatonin affect visual acuity in CSCR? Researchers will compare placebo (a look-like substance that contains no drug) to see if melatonin works to treat CSCR.

Participants will:

1. Take melatonin or placebo twice a day for one month
2. Visit the clinic after finishing a course of treatment, and 1 and 3 months after that for visual acuity assessment and tests
3. Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose diagnosis of central serous chorioretinopathy is confirmed based on clinical and imaging criteria within the past 6 weeks
2. Patients with minimum age of 18 years old
3. Consent to participate in the study

Exclusion Criteria:

1. A history of vitrectomy
2. A history of laser surgery in the eye being studied in the past 3 months
3. A history of anti-VEGF injection in the eye being studied in the past 3 months
4. History of patient suspicious for choroidal neovascularization (CNV)
5. Pregnant or nursing patients
6. Patients with significantly compromised visual acuity in the eye being studied due to concomitant ocular condition
7. Patients participating in any other investigational drug study
8. Inability to obtain OCT photographs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
central macular thickness (CMT) | From enrollment to 3 month later
  Changes in central macular thickness (CMT) in patients receiving oral melatonin versus patients receiving placebo
best visual acuity (BCVA) | From enrollment to 3 months later
  Changes in best visual acuity (BCVA) in patients receiving oral melatonin versus patients receiving placebo

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Pourazizi, Study Director — Isfahan University of Medical Sciences, Feiz Hospital, Isfahan Isfahan, Isfahan, Iran